CLINICAL TRIAL: NCT04335435
Title: Avenanthramide and Saponin Bioavailability in Oat Bran
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Shengmin Sang, Principal Investigator, North Carolina Agriculture & Technical State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-0179
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Human Health; Polyphenols; Pharmacokinetics
Keywords: Avenanthramides; Saponins; bioavailability; polyphenols; oat bran; pharmacokinetics
MeSH Terms: interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oat Bran Consumption (Experimental): Each subject consumed 120 g of oat bran (by dry weight) in a single dose, and samples (urine and fecal) were collected at different time points following the administration of oat bran.
  Interventions: Dietary Supplement: Oat Bran Consumption

INTERVENTIONS:
Dietary Supplement: Oat Bran Consumption — Oat bran (120 g), single dose.
  Other Names: Gut Microbiome and Oat metabolism Study

SUMMARY:
Avenanthramides and saponins are types of chemical compounds found naturally in oats.

Avenanthramides have anti-oxidant properties, anti-atherosclerotic, anti-inflammation, and anti-proliferative effects on cancer cells in vitro. Oat saponins, or avenacosides, have the ability to bind cholesterol, and thus, the ability to lower blood cholesterol.

Oat bran is a known source of these dietary compounds. This study aims to determine the bioavailability of these compounds to in the urine of participants after ingesting an oat bran cereal, both before, and after for multiple time points.

Analytical chemistry will be used to determine the bioavailability of the oat compounds at each time point. This will help to establish a kinetic curve for the metabolism of these compounds.

DETAILED DESCRIPTION:
Initially, the diet of the participants will be asked to restricted to avoid eating any polyphenols that might interfere with the employed analytical chemistry techniques. This period of diet restriction is the washout period. The list of foods to avoid are: oats, whole grains, fruits, vegetables, herbal supplements, ginger, coffee, tea, and chocolate.

After the washout period, a baseline urine and fecal sample will be collected from the participants, then a large portion of oat bran will be provided to the participants for consumption. The approximate portion size will be 100 g by dry weight. The participants will then provide urine samples during the designated time points. The time points for the urine collection are as follows:

1. st sample, ~ 30 min to 1 hour prior to oat consumption
2. nd sample: 0-2 hours after oat consumption
3. rd sample: 2-4 hours after oat consumption
4. th sample: 4-6 hours after oat consumption
5. th sample: 6-9 hours after oat consumption
6. th sample: 9-12 hours after oat consumption
7. th sample: 12-24 hours after oat consumption
8. th sample: 24-32 hours after oat consumption
9. th sample: 48 hours after oat consumption These samples will be analyzed in using HPLC and LC/MS.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-25
* Have blood and urine biochemical markers in normal range
* Have no known allergy to oat relate foods
* Be not taking antibiotics for six months
* Be not currently taking medication
* Be nonsmoking
* Have no alcoholic intoxication
* Have no extensive exposure to industrial waste

Exclusion Criteria:

* Individuals with gout
* Individuals with heart disease
* Individuals with peripheral vascular diseases
* Individuals with degenerative liver
* Cancer patients
* Patients with diabetes
* Individuals with GI disorders
* Individuals with endocrine disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2016-01-21 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Avenanthramides and Saponins in Urine | 0-2 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 2-4 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 4-6 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 6-9 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 9-12 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 12-24 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 24-32 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.
Bioavailability of Avenanthramides and Saponins in Urine | 32-48 hours post-dose
  Liquid chromatography-tandem mass spectrometry will be utilized to assess the bioavailability of avenanthramides and saponins in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Shengmin Sang, PhD, Principal Investigator — North Carolina Agriculture and Technical State University

REFERENCES:
- [Derived] Wang P, Zhang S, Yerke A, Ohland CL, Gharaibeh RZ, Fouladi F, Fodor AA, Jobin C, Sang S. Avenanthramide Metabotype from Whole-Grain Oat Intake is Influenced by Faecalibacterium prausnitzii in Healthy Adults. J Nutr. 2021 Jun 1;151(6):1426-1435. doi: 10.1093/jn/nxab006. PMID 33694368